CLINICAL TRIAL: NCT04218162
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Study to Evaluate Efficacy and Safety of Lasmiditan Compared to Placebo in the Acute Treatment of Migraine
Brief Title: Lasmiditan Compared to Placebo in the Acute Treatment of Migraine in Korean
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-LAS-301
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acute Migraine
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lasmiditan 50mg (Experimental)
  Interventions: Drug: Lasmiditan 50mg
- Lasmiditan 100mg (Experimental)
  Interventions: Drug: Lasmiditan 100mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan 50mg — Lasmiditan 50mg
  Arms: Lasmiditan 50mg
Drug: Lasmiditan 100mg — Lasmiditan 100mg
  Arms: Lasmiditan 100mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled parallel group study to evaluate efficacy and safety of lasmiditan tablet compared to Placebo in the acute treatment of Migraine

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male or female, aged 18 years or above.
* Participants with migraine with or without aura fulfilling the International Headache Society (IHS) diagnostic criteria 1.1 and 1.2.1 (International Headache Classification (ICHD-3).
* History of disabling migraine for at least 1 year.
* Migraine Disability Association (MIDAS) score ≥11.
* Migraine onset before the age of 50 years.
* History of 3 - 8 migraine attacks per month (< 15 headache days per month).
* Females of child-bearing potential must be using or willing to use a highly effective form of contraception (e.g. combined oral contraceptive, intrauterine device (IUD), abstinence or vasectomized partner).
* Able and willing to complete an electronic diary to record details of the migraine attack treated with study drug.

Exclusion Criteria:

* Any medical condition or clinical laboratory test which in the judgment of the Investigator makes the participant unsuitable for the study.
* Pregnant or breast-feeding women.
* Known hypersensitivity to lasmiditan or to any excipient of lasmiditan oral tablets, or any sensitivity to lasmiditan.
* History or evidence of hemorrhagic stroke, epilepsy or any other condition placing the participant at increased risk of seizures.
* History of recurrent dizziness and/or vertigo including benign paroxysmal positional vertigo (BPPV), Meniere's disease, vestibular migraine, and other vestibular disorders.
* History of diabetes mellitus with complications (diabetic retinopathy, nephropathy or neuropathy).
* History within the previous three years or current evidence of abuse of any drug, prescription or illicit, or alcohol.
* History of orthostatic hypotension with syncope.
* Significant renal or hepatic impairment.
* Participant is at imminent risk of suicide (positive response to question 4 or 5) on the Columbia-Suicide Severity Rating Scale (C-SSRS) or had a suicide attempt within six months prior to screening.
* Participation in any clinical trial of an experimental drug or device in the previous 30 days.
* Known Hepatitis B or C or human immunodeficiency virus(HIV) infection. History, within past 12 months, of chronic migraine or other forms of primary or secondary chronic headache disorder (e.g. hemicranias continua, medication overuse headache) where headache frequency is ≥15 headache days per month.
* Use of more than 3 doses per month of either opiates or barbiturates.
* Initiation of or a change in concomitant medication to reduce the frequency of migraine episodes within three (3) months prior to Screening/Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Headache Pain Free at 2 Hours Post Dose | 2 hours post dose
  The percentage of participants defined as mild, moderate, or severe headache pain becoming none.

SECONDARY OUTCOMES:
Percentage of Participants Who Are Most Bothersome Symptom (MBS) Free | 2 hours post dose
  The percentage of participants defined as the associated symptom present and identified as MBS (nausea, photophobia, or phonophobia) prior to dosing being absent.
Percentage of Participants With Headache Relief | 2 hours post dose
  The percentage of participants with headache pain moderate or severe which became mild or none or with headache pain mild which became none.
Number of Participants With Headache Recurrence | 2 Hours Post Dose Up to 48 Hours
  The number of participants with headache recurrence
Percentage of Participants Use of Rescue Medication | From 2 Hours Post Dose Up to 24 Hours
  The percentage of participants who used rescue medication.
Number of Participants With Treatment Emergent Adverse Events | From Baseline Up to End of Study
  Safety and tolerability was assessed by the number of participants with at least 1 treatment adverse emergent event.

CONTACTS AND LOCATIONS:
Locations (1):
- IlDong Pharmaceutical Co Ltd, Seoul, South Korea